CLINICAL TRIAL: NCT03189615
Title: Interventional, Open-label, Three-group, Single-dose Study Investigating the Pharmacokinetic Properties of Lu AF35700 in Subjects With Hepatic Impairment (Mild or Moderate) and in Healthy Subjects
Brief Title: Study Investigating the Pharmacokinetic Properties of the Drug Lu AF35700 in Subjects With Liver Impairment and in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17256A; 2016-004139-20 (EudraCT Number)
Record Dates: First submitted 2017-06-14; First posted 2017-06-16 (Actual); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Hepatic Impairment
MeSH Terms: interventions — Lu AF35700

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Patients with mild hepatic impairment (Group1) (Experimental)
  Interventions: Drug: Lu AF35700
- Patients with moderate hepatic impairment (Group 2) (Experimental)
  Interventions: Drug: Lu AF35700
- Healthy subjects (Group 3) (Experimental)
  Interventions: Drug: Lu AF35700

INTERVENTIONS:
Drug: Lu AF35700 — Single oral dose of 10 mg Lu AF35700

SUMMARY:
The purpose of this study is to assess the impact of mild to moderate hepatic impairment on the pharmacokinetics of a single oral dose of Lu AF35700

ELIGIBILITY:
Inclusion Criteria:

* Subjects with hepatic impairment disease stage Child-Pugh's Criteria A (mild) or Child-Pugh's Criteria B (moderate) and healthy subjects with normal hepatic function
* Subjects have a body mass index between 18.5 and 34 kg/m2 (inclusive)

Exclusion Criteria:

* Subjects previously been dosed with Lu AF35700

Other protocol defined inclusion and exclusion criteria may apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-05-14 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-04-23 (Actual)

PRIMARY OUTCOMES:
Area under the Lu AF35700 plasma concentration-time curve from zero to infinity (AUC0-inf) | Predose to day 57 postdose
  Area under the Lu AF35700 plasma concentration-time curve from zero to infinity (AUC0-inf)
Maximum observed plasma concentration (Cmax) of Lu AF35700 | Predose to day 57 postdose
  Maximum observed plasma concentration (Cmax) of Lu AF35700

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (1):
- APEX, Munich, Germany